CLINICAL TRIAL: NCT00157677
Title: Selective D-Dimer Testing Compared With Uniform D-Dimer Testing in the Diagnosis of Deep Vein Thrombosis: A Randomized Trial
Brief Title: Selective D-Dimer Testing Compared With Uniform D-Dimer Testing in the Diagnosis of Deep Vein Thrombosis (SELECT)
Acronym: SELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CTMG-2005-SELECT; Grant Number: NA 5429
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Deep Vein Thrombosis
Keywords: deep vein thrombosis; pulmonary embolism; D-dimer testing
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Selective D-Dimer use
  Interventions: Procedure: D-dimer testing
- 2 (Active Comparator): Uniform D-Dimer use
  Interventions: Procedure: D-dimer testing

INTERVENTIONS:
Procedure: D-dimer testing — Uniform D-dimer use
  Arms: 2
Procedure: D-dimer testing — Selective D-Dimer use
  Arms: 1

SUMMARY:
The purpose of this study is to compare two diagnostic interventions to improve the way D-dimer blood testing (MDA D-dimer) is used to diagnose first time symptomatic deep vein thrombosis.

DETAILED DESCRIPTION:
* Limiting use of D-dimer testing to outpatients with a Low or Moderate clinical pretest probability (C-PTP)for deep vein thrombosis AND using a D-dimer level of < 1.0 µg FEU/mL to exclude deep vein thrombosis in those with a Low C-PTP, and a D-dimer level of < 0.5 µg FEU/mL to exclude deep vein thrombosis in those with a Moderate C-PTP, is as safe and a more efficient way to diagnose DVT than:
* Performing D-dimer testing in all patients with suspected deep vein thrombosis with use of a single D-dimer value of < 0.5 µg FEU/mL to exclude thrombosis (current practice).

All randomized patients, including those who are treated for deep vein thrombosis after initial testing, will be followed for a period of 3 months to monitor for signs and symptoms suggestive of deep vein thrombosis, pulmonary embolism, bleeds and death.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Presenting with symptoms compatible with clinically suspected deep vein thrombosis

Exclusion Criteria:

* Treatment with full dose anticoagulation for 24 hours or more.
* Other test for deep vein thrombosis already performed.
* Ongoing need for therapeutic anticoagulant therapy.
* Life expectancy less than 3 months.
* Absence of acute symptoms within 7 days of presentation.
* Presenting with symptoms of pulmonary embolism.
* Previous confirmed episode of deep vein thrombosis or pulmonary embolism.
* Current pregnancy.
* Geographic inaccessibility which precludes follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1727 (Actual)
Dates: Start 2004-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
objectively confirmed proximal deep vein thrombosis or pulmonary embolism during 3 months of follow-up in patients who are not diagnosed with deep vein thrombosis during diagnostic testing and are not anticoagulated | 3 Months

SECONDARY OUTCOMES:
bleeding | 3 Months
healthcare utilization | 3 Months
cost-effectiveness | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Linkins, MD, Principal Investigator — McMaster University; Clive Kearon, MD, Principal Investigator — McMaster University; Jim Julian, MMath, Principal Investigator — McMaster University, Dept. of Clinical Epidemiology and Biostatistics
Locations (5):
- Canada (5):
  - Hamilton Health Sciences, McMaster, Hamilton, Ontario
  - St. Joseph's Health Care Centre, Hamilton, Ontario
  - Hamilton Health Sciences, Henderson, Hamilton, Ontario
  - Hamilton Health Sciences, General, Hamilton, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Linkins LA, Bates SM, Lang E, Kahn SR, Douketis JD, Julian J, Parpia S, Gross P, Weitz JI, Spencer FA, Lee AY, O'Donnell MJ, Crowther MA, Chan HH, Lim W, Schulman S, Ginsberg JS, Kearon C. Selective D-dimer testing for diagnosis of a first suspected episode of deep venous thrombosis: a randomized trial. Ann Intern Med. 2013 Jan 15;158(2):93-100. doi: 10.7326/0003-4819-158-2-201301150-00003. PMID 23318311